CLINICAL TRIAL: NCT07172776
Title: A Community Engagement Approach to Improving Communication With Black Men About Oral and Pharyngeal Cancers
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Project Brotherhood (Unknown); American Cancer Society, Inc. (Other); University of Maryland, Baltimore County (Other)
Responsible Party: Principal Investigator, Patrick Dean Smith, Associate Professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: STUDY2022-0658; CHERC-MSI-21-168-01-CHERC-MSI (Other Grant/Funding Number: American Cancer Society)
Record Dates: First submitted 2025-09-08; First posted 2025-09-15 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2025-12

CONDITIONS: Oral Cancers
Keywords: oral cancer communication
MeSH Terms: conditions — Mouth Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre-post survey (Experimental): Participants will complete a pre-survey either on paper or online, engage with a dentist or dental student, then complete a post-survey.
  Interventions: Behavioral: oral cancer communication tool

INTERVENTIONS:
Behavioral: oral cancer communication tool — The overall goal is to determine if the OPC communication tool has potential to enhance Black-men's and dentists' comfort discussing oral and pharyngeal cancers in clinical-like settings.
  Each Aim builds upon activities from the previous Aim. Aim 1a and Aim1b activities will produce a culturally- aligned oral-pharyngeal cancer communication (COPC) tool that will be used in Aim 2. In Aim 2 activities, dental providers will receive training on the tool and practice utilization of the tool. The tool will be further revised using the additional feedback from Aim 2 activities. In Aim 3, the revised culturally- aligned COPC tool will be utilized in community-based settings. In this IRB amendment-modification, we are seeking approval for Phase III/ Aim 3 activities.

SUMMARY:
1. Specific OPC patient communication (COPC) tool to address OPCs among Black men.
2. Assess the COPC tool's ability to improve dental providers' communication with Black men.
3. Implement a pilot test of the culturally tailored OPC communication tool in community-based settings to assess perceptions, knowledge and experiences of Black men receiving oral cancer screenings

DETAILED DESCRIPTION:
Aim 1: Adapt an existing OPC patient communication tool into a culturally- specific OPC patient communication (COPC) tool to address OPCs among Black men.

Aim 1a: We will use a mixed methods study design to conduct focus groups/ interviews and surveys among Black men who reside or work in UI Health catchment areas (n=25).

Aim 1b: Up to 20 Black males will be recruited by the research team to review the communication tool and infographic and participate in discussions to assess the tool's acceptability, cultural appropriateness, and potential to improve communication with Black men about OPCs. The communication tool is a document that will be used by dentists to communicate with and screen patients for OPC in culturally sensitive manner. Based on feedback from the Aim 1b focus group participants, the research team will further revise the COPC tool to ensure that it is culturally aligned, acceptable, and appropriate.

Aim 2: Assess the COPC tool's ability to improve dental providers' communication with Black men about OPCs in a simulated environment.

We will train up to 15 dental providers to use the tool (n=15). They will receive an introduction to the tool, use the tool during a simulated patient encounter and complete an interview to assess their overall attitudes of the tool, the tool's usability, and its effectiveness in helping to improve their self-efficacy for communicating with Black men about OPCs. The dental providers will complete a one-on-one individual interview. There will not be any focus groups in Aim 2 activities.

Aim 3: Implement a pilot test of the culturally tailored OPC communication tool in community-based settings to assess the perceptions, knowledge and experiences of Black men receiving oral cancer screenings.

Aim 3a) Up to 50 Black male oral cancer screening patients will be invited to complete pre surveys and post surveys to assess the tool's effectiveness in improving their OPC knowledge and comfort discussing OPCs. Oral cancer screening examinations are offered as part of the research along with the OPC Communication Tool, the OPC Infographic and the surveys. Participants have the option of NOT completing the oral cancer screening examinations but still completing the rest of the research.

Aim 3b) Up to 50 Dentists and dental students will use the OPC Communication Tool and OPC Infographic to conduct oral cancer screenings. Oral cancer screening examinations are offered as part of the research along with the OPC Communication Tool, the OPC Infographic and the surveys. Participants have the option of NOT completing the oral cancer screening examinations but still completing the rest of the research. The dentists and dental students conducting the OPC screenings will complete a demographic survey and a post survey.

ELIGIBILITY:
Aim 1a Inclusion Criteria

1) Self-Identify as African American or Black 2) Self-Identify as male 3) Age 18 and over 4) Reside or work in the UI Cancer Center catchment area Exclusion Criteria

1. Does not self-identify as African American or Black
2. Does not self-identify as male
3. Less than Age 18
4. Does not reside or work in the UI Cancer Center catchment area
5. Is a dental professional or dental student

Aim 1b Inclusion Criteria

1. Self-Identify as African American or Black
2. Self-Identify as male
3. Age 18 and over
4. Reside or work in the UI Cancer Center catchment area Exclusion Criteria

1) Does not self-identify as African American or Black 2) Does not self-identify as male 3) Less than Age 18 4) Does not reside or work in the UI Cancer Center catchment area 5) Is a dental professional or dental student Aim 2 Inclusion Criteria

1. Licensed as a general dentist in IL
2. Age 18 and over
3. Practice general dentistry in the University of Illinois Cancer Center catchment area
4. Self-reported to provide general dentistry care to at least one Black male patient per week Exclusion Criteria

<!-- -->

1. Not licensed as a general dentist in IL
2. Not Age 18 and over
3. Does not practice general dentistry in the University of Illinois Cancer Center catchment area
4. Does not self-report to provide general dentistry care to at least one Black male patient per week

Aim 3a Inclusion Criteria for Oral Cancer Screening patients 1) Self-Identify as African American or Black 2) Self-Identify as male 3) Age 18 and over 4) Reside or work in the UI Cancer Center catchment area Exclusion Criteria for Oral Cancer Screening patients

1. Does not self-identify as African American or Black
2. Does not self-identify as male
3. Less than Age 18
4. Dentists and/ or Dental Students

Aim 3b Inclusion Criteria for Dentists and/or Dental students

1. Licensed as a general dentist or legally able to provide dental screenings under the direct supervision of a dentist licensed in Illinois
2. Age 18 and over
3. Practice general dentistry in the University of Illinois Cancer Center catchment area
4. Dental students must be either a third or fourth year dental student enrolled at UIC College of Dentistry Exclusion Criteria for Dentists and/or Dental students

1) Not licensed as a general dentist in IL or is not legally able to provide dental screenings under the direct supervision of dentist licensed in Illinois 2) Not Age 18 and over 3) Does not practice general dentistry in the University of Illinois Cancer Center catchment area 4) Dental students must not be at a level below that of a third or fourth year dental student enrolled at UIC College of Dentistry

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Male
Enrollment: 50 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
oral cancer communication | 10 minutes
  This communication tool will ideally help dentists communicate with their patients about oral cancer risk and treatment. The oral cancer screenings will occur in person. Participants will complete a pre-survey either on paper or online, engage with a dentist or dental student, then complete a post-survey

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Smith PD, Murray M, Bailey T, Peterson CE, Bekoe O, Weatherspoon DJ. A community-based participatory protocol to improving communication with Black men about oral and pharyngeal cancers: Research protocol. PLoS One. 2023 Aug 17;18(8):e0288478. doi: 10.1371/journal.pone.0288478. eCollection 2023. PMID 37590209